CLINICAL TRIAL: NCT03433326
Title: A Multicenter, Open Label, Pilot Study of MK-5172 (Grazoprevir)/MK-8742 (Elbasvir) Without Ribavirin for 12 Weeks in G1b and G4 Patients With HCV-related Cryoglobulinemic Nephropathy
Brief Title: Grazoprevir and Elbasvir Without Ribavirin for 12 Weeks in Patients With HCV-related Cryoglobulinemic Nephropathy
Acronym: CRYOKID
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Florence (Other)
Responsible Party: Principal Investigator, Anna Linda Zignego, professor of internal medicine, University of Florence
Other Study IDs: 56086
Record Dates: First submitted 2018-02-08; First posted 2018-02-14 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Hepatitis C; Cryoglobulinaemic Glomerulonephritis
MeSH Terms: conditions — Hepatitis C | interventions — elbasvir-grazoprevir drug combination

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Weeks
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Elbasvir/Grazoprevir — Administration of MK-8742 (Elbasvir)/MK-5172 (Grazoprevir) for 12 weeks
  Other Names: MK-8742/MK-5172

SUMMARY:
CryoKid is a no-profit, multi-center, single-arm, open-label, pilot study. The study aims to evaluate the tolerability of MK-8742 (Elbasvir) / MK-5172 (Grazoprevir) administrated for 12 weeks without Ribavirin in patients with HCV chronic hepatitis (G1b and G4) and cryoglobulinemic nephropathy.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent form signed,
2. Male or female at least 18 years of age at time of Screening.
3. Chronic infection with Hepatitis C virus G1b
4. Chronic infection with Hepatitis C virus G4 naïve, and experienced with baseline HCV RNA level <800,000 IU/ml
5. Metavir score ranging between F0-F4 (with Child-Pugh score ranging from A5 to A6)
6. Diagnosis of mixed cryoglobulinemia MC (type III or II) according to standard criteria
7. Chronic renal impairment due to cryoglobulinemic nephropathy. Subjects with renal impairment will include CKD Stage 5 (eGFR < 15mL/min or dialysis dependent), CKD Stage 4 (eGFR 15-29 mL/min), CKD Stage 3 eGFR (30-59 mL/min) and CKD Stage 2 (60-89 mL/min) HCV patients.
8. Albumin level ≥ 3.0 g/dl,
9. Platelet count ≥ 75 x 103/μL.

Exclusion Criteria:

1. Age <18 years
2. Chronic infection with Hepatitis C virus G4 experienced with baseline HCV RNA level >800,000 IU/ml
3. Patients with HCV genotype 1a, 2, 3, 5, 6,
4. Coexistence of life-threatening condition(s) unrelated to MC
5. Diagnosis of malignancy
6. Pregnancy or breast feeding.
7. Child-Pugh score > A6
8. Decompensated cirrhosis or previous decompensation
9. Platelet count < 75 x 103/μL
10. Albumin level < 3 g/l
11. Co-infection with more than one HCV genotype.
12. Any serious or active medical illness which, in the opinion of the investigator, would interfere with subject treatment, assessment, or compliance
13. HIV or chronic hepatitis B virus (HBV) infection (HBsAg positive)
14. Known hypersensitivity to Grazoprevir, Elbasvir or any of its components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: G1b and G4 patients with HCV-related Cryoglobulinemic Nephropathy
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
SVR12 | march 2018-october 2018
  Percentage of participants achieving sustained virologic response 12 weeks after completing treatment (SVR12)

SECONDARY OUTCOMES:
SVR24 | march 2018-december 2018
  Percentage of participants achieving Sustained Virologic Response 24 weeks after ending study treatment (SVR 24)
Clinical response: improvement or disappearance of MC clinical and biochemical stigmata | march 2018-december 2018
  Clinical response: improvement or disappearance of MC clinical and biochemical stigmata at the EOT, at week 12 and week 24 of follow-up. Improvement of the renal function at week 4, week 8, EOT at week 12 and week 24 of follow-up.
Tolerability: Number of participants experiencing an adverse event (AE) | march 2018-may 2018
  Tolerability: Number of participants experiencing an adverse event (AE)

CONTACTS AND LOCATIONS:
Overall Officials: ANNA LINDA ZIGNEGO, MD, PhD, Principal Investigator — University of Florence

IPD SHARING:
Plan to Share IPD: No